CLINICAL TRIAL: NCT04606979
Title: The Potential of Transcranial Direct Current Stimulation of the Primary Motor Cortex to Promote Implicit Motor Sequence Learning in Individuals With Parkinson's Disease and Age-matched Healthy Controls
Brief Title: tDCS of the Primary Motor Cortex to Improve Implicit Motor Sequence Learning in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Mahyar Firouzi, Principle Investigator (Doctoral Researcher), Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B1432020000012
Record Dates: First submitted 2020-10-10; First posted 2020-10-28 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease; Parkinson; Healthy
Keywords: Parkinson Disease; Transcranial Direct Current Stimulation; tDCS; Serial Reaction Time Task; Sequence Learning; Procedural Learning; Implicit Learning; Implicit Motor Sequence Learning
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: sham-controlled, counterbalanced study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parkinson Disease - Group 1a - Active tDCS first (Experimental): Half of the subjects with PD will receive active (anodal, real) tDCS in the first session. Following cross-over and a three-week washout-period, this half of the subjects with PD will receive sham (placebo) tDCS.
  Interventions: Device: 1x1 Low Intensity Transcranial Direct Current Stimulation (tDCS)
- Parkinson Disease - Group 1b - Sham tDCS first (Sham Comparator): Half of the subjects with PD will receive sham tDCS in the first session. Following cross-over and a three-week washout-period, this half of the subjects with PD will receive active (anodal, real) tDCS.
  Interventions: Device: 1x1 Low Intensity Transcranial Direct Current Stimulation (tDCS)
- Healthy Controls - Group 2a - Active tDCS first (Experimental): Half of the healthy controls will receive active (anodal, real) tDCS in the first session. Following cross-over and a three-week washout-period, this half of the healthy controls will receive sham (placebo) tDCS.
  Interventions: Device: 1x1 Low Intensity Transcranial Direct Current Stimulation (tDCS)
- Healthy Controls - Group 2b - Sham tDCS first (Sham Comparator): Half of the healthy controls will receive sham tDCS in the first session. Following cross-over and a three-week washout-period, this half of the healthy controls will receive active (anodal, real) tDCS.
  Interventions: Device: 1x1 Low Intensity Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: 1x1 Low Intensity Transcranial Direct Current Stimulation (tDCS) — tDCS will be delivered through a pair of identical square rubber electrodes (size 35 cm2), placed in rectangular saline-soaked sponges. For the stimulation of M1, electrodes will be placed over C3 or C4 according to the 10-20 EEG system, matching with the M1 contralateral to the performing dominant hand. The reference electrode will be positioned on F1 or F2, ipsilateral to the dominant hand.
  The current stimulation will be slowly ramped up from 0 mA to 2 mA in one minute. For the anodal tDCS condition, this intensity will be maintained for the duration of the SRT-task (approximately 20 minutes). This will result in a current density of 0,057 mA/cm2. For the sham tDCS condition - unbeknown to the subject - stimulation will be gradually decreased towards 0 mA immediately after the one-minute ramp-up. During the last block of the SRT-task, this gradual ramping-up and -down of the current stimulation will be repeated to optimize the process of blinding of participants.

SUMMARY:
Implicit motor sequence learning (IMSL) is a form of cognitive function that is known to be directly associated with impaired motor function in Parkinson's disease (PD). Research in healthy young participants shows the potential for transcranial direct current stimulation (tDCS), a non-invasive brain stimulation technique, over the primary motor cortex (M1) to enhance IMSL. tDCS has direct effects on the underlying cortex, but also induces distant (basal ganglia) network effects - hence its potential value in PD, a prime model of basal ganglia dysfunction. To date, however, only null-effects have been reported in persons with PD. In the present study, the investigators will investigate the potential of tDCS delivered over M1 to enhance IMSL, as measured by the Serial Reaction Time task, in persons with PD. The investigators will determine immediate effects that may occur concurrently with the application of tDCS but also short-term (five minutes post-tDCS) and long-term (one week post-tDCS) consolidation effects, as previous studies suggest that tDCS exerts its beneficial effects on IMSL in a consolidation phase rather than in an acquisition phase. Establishing possible consolidation effects is of a particular interest, as long-term effects are vital for the successful functional rehabilitation of persons with PD.

DETAILED DESCRIPTION:
STUDY DESIGN

The investigators will conduct a single-blind, sham-controlled, counterbalanced study to investigate the effects of M1 tDCS on IMSL. As age-related effects may serve as an explanation for the conflicting findings in healthy young adults and persons with PD, the investigators will include a healthy control group, age-matched to the PD group. For the sequence-specific aspect of IMSL (primary outcome), a mixed factorial repeated measures ANOVA will be carried out with "group" (2 levels: PD, healthy) as between-subjects factor and "stimulation" (2 levels: anodal, sham), "blocks" (2 levels: random block, mean of adjacent blocks) and "time" (3 levels: during, post5min, post1week) as within-subjects factors. Similarly, for general learning (secondary outcome), a mixed factorial repeated measures ANOVA will be carried out with "group" (2 levels: PD, healthy) as between-subjects factor and "stimulation" (2 levels: anodal, sham), "blocks" (7 levels: Blocks 1-6, Block 8) and "time" (3 levels: during, post5min, post1week) as within-subjects factors. All participants will receive both anodal (real) and sham (placebo) tDCS in a random order. Counterbalancing will be done by an independent investigator using Microsoft Excel®. Baseline scores on the Scales for Outcomes in Parkinson's disease COGnition (SCOPA-COG), Montreal Cognitive Assessment (MoCA) and Hospital Anxiety and Depression Scale (HADS) questionnaires, as well as clinical subtypes (akinetic-rigid subtype, tremor subtype) and sequence awareness scores will be taken up as covariates.

RECRUITMENT STRATEGY

Persons with PD will be recruited via following instances and centres: the Flemish Parkinson Liga (VPL); neurologists of the University Hospital of Brussels (UZ Brussel), University Colleges Leuven-Limburg (UCLL) and RevArte rehabilitation centre (Antwerp); private physiotherapy practitioners specialized in neurologic rehabilitation. Age-matched healthy participants will be recruited via the PD candidates (partners of the patients), several residential care homes in and around Brussels and by posting digital flyers on social media.

There are no restrictions or prohibitions for the subjects. Participants will continue to take their medication during the trial period, and will perform the experimental procedure during the ON-phase of their medication. This is in order to maximize feasibility to perform the task and for the sake of uniformity with previous studies examining tDCS effects in PD.

MATERIALS

A 1x1 Low Intensity Direct Current Stimulator (Soterix Medical Inc, New York, USA) will be used to generate and deliver tDCS through a pair of identical square rubber electrodes (size 35 cm2), placed in rectangular saline-soaked sponges. For the stimulation of M1, electrodes will be placed over C3 or C4 according to the international 10-20 electroencephalogram system, matching with the M1 contralateral to the performing hand. The reference electrode will be positioned on F1 or F2, ipsilateral to the performing hand.

The current stimulation will be slowly ramped up from 0 milliampere (mA) to 2 mA in one minute. For the anodal tDCS condition, this intensity will be maintained for the duration of the SRT-task (approximately 20 minutes), which is well within evidence-based safety standards for tDCS. This will result in a current density of 0,057 mA/cm2. For the sham tDCS condition - unbeknown to the subject - stimulation will be gradually decreased towards 0 mA immediately after the one-minute ramp-up. During the last block of the SRT-task, this gradual ramping-up and -down of the current stimulation will be repeated to optimize the process of blinding of participants. To control for blinding of the subjects, after the last session subjects will be asked whether they were aware of the stimulation condition or not. Transient side-effects will be inventoried by the experimenter during and two weeks after the tDCS protocol, including a slight itching sensation under the electrode, redness of the skin under the electrode, headache, nausea, fatigue or insomnia.

The Serial Reaction Time task (SRT-task) will be used to determine IMSL. The SRT- task will be performed on a laptop using E-Prime® software (Psychology Software Tools, Inc., Pittsburgh, Pennsylvania, USA). Participants will be asked to press the horizontally aligned response keys C, V, B, N of a standard azerty keyboard for a leftmost, left, right, rightmost target, respectively. Responses will be given with the index finger of the least affected hand in the case of the persons with PD and with the dominant hand in the case of the healthy controls. If both hands are equally affected in the persons with PD, the dominant hand will be used as well. The response keys C, V, B and N will be the only visible keys, all other keys will be covered.

PROCEDURE

The experiment will take place at a laboratory of the Vrije Universiteit Brussel (VUB), in the participants' home environment, or at a nearby community centre of their choosing, under supervision of the investigator. The option to conduct the experiment outside of our laboratory at the VUB is given as displacements are not always evident for these participants.

The experimental procedure will be preceded by an in-person interview to collect general clinical and demographic characteristics. A shortened, 3-block x 25 trials random SRT-task will also be performed to assess whether participants have sufficient motor function to complete the experiments. Following the interview, a neuropsychological assessment will be done by means of three questionnaires:

* The Montreal Cognitive Assessment (MoCA) will be used to assess cognitive function across 8 domains (executive functions, visuospatial skills, attention, concentration, language, short term memory and orientation).
* The Scales for Outcomes in Parkinson's disease, COGnition part (SCOPA-COG) is a short, reliable and valid instrument for the assessment of cognitive function in PD. It consists of 10 items, divided over four domains: memory (4 items), executive function (3 items), attention (2 items) and visuospatial function (1 item). Scored 0-43, with lower scores indicating more severe cognitive impairment.
* The Hospital Anxiety and Depression Scale (HADS) is a two-dimension scale developed to identify depression and anxiety. It consists of 14 items, divided into two 7-item subscales. Each item is rated on a 4-point scale ranging from 0 (absence) to 3 (extreme presence).

Furthermore, participants' motor function will be assessed by means of:

• The Unified Parkinson's Disease Rating Scale, part III (UPDRS-III), one of the most widely used clinical rating scales for PD, which consists of 4 parts. For the present study, only part III will be used, which assesses motor function by means of 14 items.

Following the screening session (T0), all eligible participants will be seen four times (T1-T4) over the course of minimally five to maximally eleven weeks. All four sessions (T1, T2, T3, T4) will start with a practice block of the SRT-task consisting of 72 random trials, followed by the actual experimental SRT-task of eight blocks of 72 trials. Blocks will be separated by a thirty second break. In Blocks 1 through 6 and Block 8, the order of the target (i.e. black dot) locations will follow a repeating sequence. This is unbeknown to the participant. The rationale is that reaction times will decrease with repetition of the sequence throughout blocks 1-6 and 8, denoting a general training effect (secondary outcome measure IMSL). When the sequence suddenly changes to a random sequence in Block 7, reaction time will increase in Block 7 and decrease once more in regularly sequenced Block 8, denoting a sequence-specific learning effect (primary outcome measure IMSL). To control for possible carry-over effects, the SRT-task will follow a different sequence in each stimulation condition (e.g. 132342134142 in T1-T2 and 243413241213 in T3-T4). To make sure IMSL is independent of a specific sequence, six different, structurally identical, sequences of 12 elements long will be counterbalanced between the participants.

The first interventional session (T1) will be planned at least 1 week after the screening session (T0) and will consist of active (anodal) tDCS or sham (placebo) tDCS administered during the SRT-task. Five minutes post-tDCS, subjects will be asked to carry out a short, three-block version of the SRT-task without application of tDCS to investigate potential short-term consolidation effects: Blocks 1 and 3 following the same regular sequence as earlier; Block 2 following a random sequence.

The second session (T2) will be planned one week later. During this one-week post-tDCS session the same, full version of the SRT-task from one week earlier will be performed, this time without the application of tDCS, to determine potential long-term consolidation effects. After T2, a washout period of at least three weeks will be planned to control for carry-over effects between the two stimulation conditions (active/sham tDCS). Cross-over will take place and the same procedure with the opposite stimulation condition will be repeated during the third (T3) interventional and fourth (T4) follow-up session. Half of participants in each group will have received active tDCS during T1 and sham tDCS during T3, while the other half of participants will have received these conditions in reversed and randomized order.

Each session, the SRT-task will be started within 90 minutes after medication intake ("ON-phase of medication"). This is in order to maximize feasibility to perform the task and for the sake of uniformity with previous studies examining tDCS effects in PD. A post-SRT-task questionnaire will be completed after the last session (T4) to determine whether participants became aware of the sequential nature of the task. If participants indicate that they believe a specific sequence appeared, they will have to reproduce the sequence of the last session as correct as possible. This sequential score (x/12, based on the highest number of sequence elements they can reproduce in the correct order) will serve as the outcome measure for explicit knowledge regarding the repeating sequences.

STATISTICAL ANALYSES

All statistical analyses will be carried out using International Business Machines (IBM) Statistical Package for the Social Sciences (SPSS) Statistics version 26. The level of significance will be set at α = 0.05. A trend towards significance will be defined as 0.05 ≤ α < 0.10. Bonferroni corrections for multiple comparisons will be made when necessary. Cohen's f effect sizes will be reported, with values of .10, .25, and .40 representing small, medium, and large effect sizes, respectively.

In the event of null-effects, the investigators will conclude that there is no evidence of a difference between conditions. However, the investigators will also calculate post-hoc Bayes factors for each group (PD, healthy controls) to assess whether a lack of difference in sequence learning between the anodal and sham stimulation conditions could be interpreted as evidence for the absence of an effect of tDCS on sequence learning.

For the PD group, patients will be classified as akinetic-rigid subtype or tremor subtype based on UPDRS-III subscores in the "Off" medication state. This clinical subtype of the persons with PD will be taken up as covariate, to assess whether this characteristic influences IMSL or the treatment thereof via tDCS. A method similar to the one used by Xu et al. (2018) will be used [70]. First, "tremor score" (sum of UPDRS items 20 and 21 divided by 7) and "non-tremor score" (sum of UPDRS items 18, 19, 22, 27, 28, 29, 30 and 31 divided by 12) will be calculated per patient. If the tremor score is at least twice the non-tremor score, patients are classified as tremor subtype; if the non-tremor score is at least twice the tremor score, patients are classified as akinetic-rigid subtype.

Correlation analyses, Bonferroni-corrected for multiple comparisons, will be performed to investigate if the amount of IMSL correlates with demographical, neuropsychological and clinical variables (including clinical subtypes of PD). If assumptions for parametrical testing are violated, the non-parametric alternative Spearman's Rho will be calculated.

The analyses of the SRT-task performance will be based on median reaction time (RT) per block instead of mean RT to minimize potential outlier effects. Practice trials, the first response after each break, erroneous responses and responses following an error will be excluded from the analyses. Median RTs per block will be analyzed to determine (1) a general learning effect (secondary outcome measure) and (2) a sequence-specific learning effect (primary outcome measure).

General learning effects during and one-week post-tDCS will be derived from a decline in median RTs over the seven regularly sequenced blocks (i.e. Blocks 1-6 and Block 8). This will not be applicable to the 5-minutes post-tDCS SRT-task as it is a short version with only three blocks. A 2x2x2x7 repeated measures ANOVA will be carried out with group (PD, healthy controls) as between-subjects factor and stimulation (active, sham), time (during, post1week) and block (Blocks 1-6, Block 8) as within-subjects factors.

Sequence-specific learning effects during, 5 minutes and 1 week post-tDCS will be analyzed by subtracting the mean of the median RTs of adjacent sequenced blocks (Blocks 6 and 8 during stimulation and at 1 week post-tDCS; Blocks 1 and 3 at 5 minutes post-tDCS) from the median RT of the random block (Block 7 during stimulation and at 1-week post-tDCS; Block 2 at 5-minutes post-tDCS). A 2x2x2x3 repeated measures ANOVA (or Friedman and Wilcoxon signed rank tests as non-parametrical alternatives) will be carried out with group (PD, healthy controls) as between-subjects factor and stimulation (active, sham), sequence (random block, mean of adjacent sequenced blocks) and time (during, post5min, post1week) as within-subject factors.

In case assumptions of sphericity are violated, Greenhouse-Geisser or Huynh-Feldt corrections will be reported. Bonferroni-corrected t-tests will be implemented to further analyze significant main and interaction effects.

Error percentages in the SRT-task are generally small and thus, because of a limited number of observations, less sensitive to IMSL. The percentage erroneous reactions per block will be calculated for both stimulation conditions (anodal, sham) and for the three measurements over time (concurrent, post5minutes, post1week). The Shapiro-Wilk test of residuals will be carried out to evaluate normality of distribution.

The sequential score, as outcome measure for explicit knowledge, will be taken up as a covariate in the analyses. An independent samples t-test (or non-parametrical alternative Mann-Whitney U test) will be carried out to ascertain whether the sequential scores (x/12) of the PD group are different from the healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with the idiopathic form of PD by a neurologist (PD subjects only)
* Dutch or French speaking
* sufficient upper limb motor skills to perform the SRT-task (determined by means of a practice version of the SRT-task consisting of one block of 50 random trials)
* able to signal pain or discomfort
* able to give informed consent

Exclusion Criteria:

* additional neurological disorders
* any of the following tDCS contra-indications: deep brain stimulator; pacemaker; head wound; skin condition of the scalp; a history of epilepsy

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-11 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Serial Reaction Time task: Sequence-Specific Learning Effect (during and following active tDCS) | Changes in Sequence-Specific Learning Effect will be assessed between: (baseline) during active tDCS; (short-term) 5-minutes post active tDCS; (long-term) 1 week post active tDCS
  The Serial Reaction Time task (SRT-task) will be employed, using E-Prime® software. In a typical SRT task, a target (e.g. black dot) is presented in one of four horizontal locations on a computer screen. Participants are asked to react to the target location by pressing a spatially compatible response key. They are not informed that the order of target locations follows a sequence predetermined by the experimenter. Participants are trained on the sequence in several blocks of trials, e.g.: 7 blocks of 100 trials. Typically, reaction times (RTs) decrease with practice, which is referred to as a general learning effect and constitutes the non-sequence-specific learning component of IMSL. Crucially, RTs increase when the sequence is inconspicuously replaced by a random sequence and decrease again when the predetermined sequence is reintroduced. The latter is referred to as the sequence-specific learning effect and is calculated by subtracting the mean RTs of the adjacent sequel blocks.
Serial Reaction Time task: Sequence-Specific Learning Effect (during and following sham tDCS) | Changes in Sequence-Specific Learning Effect will be assessed between: (baseline) during sham tDCS; (short-term) 5-minutes post sham tDCS; (long-term) 1 week post sham tDCS
  The Serial Reaction Time task (SRT-task) will be employed, using E-Prime® software. In a typical SRT task, a target (e.g. black dot) is presented in one of four horizontal locations on a computer screen. Participants are asked to react to the target location by pressing a spatially compatible response key. They are not informed that the order of target locations follows a sequence predetermined by the experimenter. Participants are trained on the sequence in several blocks of trials, e.g.: 7 blocks of 100 trials. Typically, reaction times (RTs) decrease with practice, which is referred to as a general learning effect and constitutes the non-sequence-specific learning component of IMSL. Crucially, RTs increase when the sequence is inconspicuously replaced by a random sequence and decrease again when the predetermined sequence is reintroduced. The latter is referred to as the sequence-specific learning effect and is calculated by subtracting the mean RTs of the adjacent sequel blocks.

SECONDARY OUTCOMES:
Serial Reaction Time task: General Learning Effect (during and following active tDCS) | Changes in General Learning Effect will be assessed between: (baseline) during active tDCS; (short-term) 5-minutes post active tDCS; (long-term) 1 week post active tDCS
  The Serial Reaction Time task (SRT-task) will be employed, using E-Prime® software. In the SRT-task, typically, reaction times (RTs) decrease with practice, which is referred to as a general learning effect and constitutes the non-sequence-specific learning component of IMSL.
Serial Reaction Time task: General Learning Effect (during and following sham tDCS) | Changes in General Learning Effect will be assessed between: (baseline) during sham tDCS; (short-term) 5-minutes post sham tDCS; (long-term) 1 week post sham tDCS
  The Serial Reaction Time task (SRT-task) will be employed, using E-Prime® software. The SRT- task will be performed on a laptop using E-Prime® software. In the SRT-task, typically, reaction times (RTs) decrease with practice, which is referred to as a general learning effect and constitutes the non-sequence-specific learning component of IMSL.

CONTACTS AND LOCATIONS:
Overall Officials: Natacha Deroost, PhD, Study Director — Vrije Universiteit Brussel - Brain Body and Cognition Research Group; Kris Baetens, PhD, Study Chair — Vrije Universiteit Brussel - Brain Body and Cognition Research Group; Chris Baeken, PhD, MD, Study Chair — University Ghent; Frank Van Overwalle, PhD, Study Chair — Vrije Universiteit Brussel - Brain Body and Cognition Research Group; Eva Swinnen, PhD, Study Chair — Vrije Universiteit Brussel - Rehabilitation Research Group; Mahyar Firouzi, PhD, Principal Investigator — Vrije Universiteit Brussel - Brain Body and Cognition Research Group
Locations (1):
- Vrije Universiteit Brussel, Brussels, Brussels Capital, Belgium